CLINICAL TRIAL: NCT03008083
Title: A Prospective Multi-center Open-label Controlled Trial of Comparison 3 vs 12 Months of Dual Anti-Platelet Therapy After Implantation of Firehawk Sirolimus Target- Eluting Stent in Patients With Stable Coronary Artery Disease
Brief Title: Comparison Three vs Twelve Months of Dual Anti-Platelet Therapy After Stent Implantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGET DAPT
Record Dates: First submitted 2016-12-06; First posted 2017-01-02 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Drug-Eluting Stents; Percutaneous Coronary Intervention
MeSH Terms: interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months DAPT Intervention (Active Comparator): After implantation of Firehawk coronary stents, all subjects in intervention group will be given dual anti-platelet therapy (DAPT) including aspirin and thienopyridines (clopidogrel or ticagrelor)for 3 months.
  Interventions: Drug: 3 months DAPT
- 12 months DAPT Intervention (Active Comparator): After implantation of Firehawk coronary stents, all subjects in control group will be given dual anti-platelet therapy (DAPT) including aspirin and thienopyridines (clopidogrel or ticagrelor)for 12 months.
  Interventions: Drug: 12 months DAPT

INTERVENTIONS:
Drug: 3 months DAPT — Subjects will continue DAPT with P2Y12 inhibitors and Aspirin (ASA) up to 90 days, after which patients will continue on monotherapy with ASA only, unless contraindications for ASA emerge.
  Other Names: Ticagrelor (180 mg/day) or Clopidogrel (75 mg/day)
  Arms: 3 months DAPT Intervention
Drug: 12 months DAPT — Subjects will continue DAPT with P2Y12 inhibitors and Aspirin (ASA) up to 360 days, after which patients will continue on monotherapy with ASA only, unless contraindications for ASA emerge.
  Other Names: Ticagrelor (180 mg/day) or Clopidogrel (75 mg/day)
  Arms: 12 months DAPT Intervention

SUMMARY:
This study is a prospective,multi-center, open-label, randomized controlled clinical trial,aims to assess the clinical noninferiority of 3 months (short-term) vs 12 months (long-term) of Dual Anti-Platelet Therapy (DAPT) in patients undergoing percutaneous coronary intervention implanted sirolimus target- eluting stent with abluminal grooves containing a biodegradable polymer (Firehawk™ stent). All participants met the inclusion criteria begin taking aspirin and open-label thienopyridine therapy before index procedure, and will be 1:1 randomized to 3 months or 12 month of DAPT at index procedure.

DETAILED DESCRIPTION:
This study will recruit 2,446 subjects with stable coronary artery disease in no more than 40 research centers in China. All participants met the inclusion criteria will be 1:1 randomized to 3 months or 12 month of DAPT after implanting Firehawk™ coronary stent.Clinical follow-up will be carried out at 30 days, 3 months, 6 months, 12 months, 18 months, 2 years and 3 years after index procedure.The primary study endpoint is Net Adverse Clinical and Cerebral Events (NACCE), a composite of all-cause death, myocardial infarction (MI), cerebral vascular accident (CVA) and major bleeding (academic research consortium [ARC] definition and GUSTO definition) at 18 months. Subjects that complete of 18 months follow-up will be regarded as having completed the primary endpoint. The secondary study endpoints contain ARC defined stent thrombosis (ST) at all study time-points; NACCE at 30 days,6,12,24 and 36 months of follow-up;major adverse cardiovascular events (MACE),major adverse cardiovascular and cerebral events (MACCE),target lesion revascularization (TLR),target lesion failure(TLF),ST at 30 days,6,12 ,18,24 and 36 months of follow-up; major bleeding at 1, 3, 6, 12 ,18,24 and 36 months of follow up; as well as cost-effective at 18 months of follow-up.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥ 18 years;
* Subjects (or legal guardians) understand the testing requirements and procedures, and provide written informed consent;
* Subjects with symptomatic coronary artery disease or confirmed asymptomatic ischemia;
* Target lesion should be new lesion with visually estimated reference diameter ≥2.5 mm and ≤4.0 mm in autologous coronary artery;
* Subjects willing to accept PCI therapy and to implant Firehawk™ stent only;
* Left ventricular ejection fraction (LVEF) ≥ 30%;
* Subjects willing to accept the trial plan calls for all subsequent evaluations.

Angiographic Inclusion Criteria:

* Target lesions must be new and have a visually estimated reference diameter ≥2.5 mm and ≤4.0 mm in autologous coronary artery;
* No limitations in target lesion length and number;
* The first target lesion must be able to successfully expand and implant Firehawk™ stent.

Clinical Exclusion Criteria:

* Subjects with ST-segment elevation myocardial infarction:
* Subjects having an organ transplant or waiting for an organ transplant
* Subjects receiving chemotherapy or going to receive a chemotherapy within 30 days after PCI
* Subjects undergoing chronic (over 72 hours) anticoagulant therapy (such as heparin and coumarin) other than acute coronary syndrome
* Subjects with abnormal counts of platelet and white blood cell (WBC) (investigator assess clinical significance combine normal reference range of laboratory)
* Subjects with confirmed or suspected liver disease, including hepatitis lab results
* Subjects with elevated serum creatinine level >3.0mg/dL or undergoing dialysis therapy
* Subjects with active peptic ulcer, active gastrointestinal (GI) bleeding or other bleeding diathesis or coagulopathy, or refused a blood transfusion
* Subjects with cerebral vascular accident (CVA) or transient ischemic attack (TIA) in the past 6 months, or with permanent nerve defects
* Subjects undergoing any PCI treatment in target vessels within 12 months prior to baseline
* Subjects planned to undergo PCI or CABG within 18 months after the baseline PCI
* Subjects with a history of any coronary endovascular brachytherapy treatment previously
* Subjects associated with drugs allergy (such as sirolimus, or structure-related compounds fluorinated polymers, thienopyridine or aspirin)
* Subjects being suffered from other serious illness (such as cancer, congestive heart failure), which may cause drop in life expectancy to less than 18 months
* Subjects with a history of drug abuse (such as alcohol, cocaine, heroin, etc.)
* Subject planned to undergo any operations that may lead to confuse with the programme
* Subjects participating in another study of drug or medical device which did not meet its primary endpoint
* Subjects planned to pregnant within 18 months after baseline
* Pregnant or breastfeeding women

Angiographic Exclusion Criteria:

* Target lesions with the following criteria: left main, saphenous vein grafts or arterial grafts, via saphenous vein grafts or arterial graft, and in-stent restenosis;
* Subjects with unprotected left main coronary artery disease (diameter stenosis >50%);
* Protected left main coronary artery disease(diameter stenosis >50% and undergoing CABG)with target lesions located in left anterior descending artery and left circumflex artery;
* Additional lesions of clinical significance possibly needing interventional within 18 months after enrollment..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2446 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical and Cerebral Events (NACCE) | At 18 months after index procedure
  A composite of all-cause death, MI, cerebral vascular accident (CVA) and major bleeding at 18 months

SECONDARY OUTCOMES:
Cost-Effectiveness Ratio (CER) | At 18 months after index procedure
  CER = [total medical care costs of anti-platelet therapy] / [number of participants without net adverse clinical and cerebral events (NACCE)]

OTHER OUTCOMES:
Net Adverse Clinical and Cerebral Events (NACCE) | In hospital and at 30 days, 3, 6, 12, 24 and 36 months after index procedure.
Major Adverse Cardiac and Cerebral Events (MACCE) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Stent Thrombosis (per ARC definition) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
  the definite and probable stent thrombosis
Target Vessel Revascularization (TVR) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Target Lesion Revascularization (TLR) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Target Vessel Failure (TVF) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Target Lesion Failure (TLF) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Myocardial Infarction (MI,including Q-wave MI and non Q-wave MI) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Major bleeding (ARC definition and GUSTO definition) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Death (All cause, Cardiac, Non-cardiac) | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Cardiac Death/ All Myocardial Infarction | In hospital and at 30 days, 3, 6, 12 ,18, 24 and 36 months after index procedure.
Procedural Success | At time of procedure up to 7 days in hospital
Minimal Lumen Diameter (MLD)（In-device, in-segment, proximal 5 mm and distal 5 mm) | Instantly after index procedure
The Immediate Lumen Gain | Instantly after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Principal Investigator — Affiliated Zhongshan Hospital of Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared. Additionally, study protocol will be available. The data will become available for the beginning 3 months and ending 5 years following article publication. The access criteria are as follow:
  * (With) Researchers who provide a methodologically sound proposal.
  * (For the analysis) to achieve aims in the approved proposal.
  * (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).
  If the data sharing plan changes after registration, this should be reflected in the statement submitted and published with the manuscript, and updated in the registry record.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: * (With) Researchers who provide a methodologically sound proposal.
  * (For the analysis) to achieve aims in the approved proposal.
  * (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Derived] Yang H, Zhang F, Zhang X, Wu Y, Zhong Z, Wang J, Zhou Y, Hong L, Yang W, Jiang T, Zou J, Zhang Z, Ma Y, Wen S, Fan Z, Xu D, Jiang H, Tao J, Ren H, Xia Y, Huang Y, Xu G, Cao R, Zheng M, Qian J, Francese DP, Lansky AJ, Ge J; TARGET DAPT Investigators. Three vs 12-month DAPT after implantation of biodegradable-polymer sirolimus-eluting coronary stent: a randomised clinical trial. BMC Med. 2025 Dec 24;23(1):690. doi: 10.1186/s12916-025-04515-y. PMID 41444578
- [Derived] Yang H, Zhang F, Yang J, Zheng M, Cao R, Dai Y, Li C, Yao K, Qian J, Ge J; TARGET DAPT trial investigators. Prospective multicentre open-label randomised controlled trial of 3-month versus 12-month dual antiplatelet therapy after implantation of the new generation biodegradable polymer sirolimus TARGET-eluting coronary stent: protocol of the TARGET DAPT trial. BMJ Open. 2019 Dec 17;9(12):e033774. doi: 10.1136/bmjopen-2019-033774. PMID 31852711